CLINICAL TRIAL: NCT01087762
Title: Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy and Safety of Certolizumab Pegol in Subjects With Active Axial Spondyloarthritis
Brief Title: Certolizumab Pegol in Subjects With Active Axial Spondyloarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS001; 2009-011719-19 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2016-11

CONDITIONS: Spondyloarthropathies
Keywords: Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Spondylarthropathies | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- CZP 200 mg Q2W (Experimental): Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 onwards.
  At every visit, subjects received one injection of 200 mg CZP and one injection of Placebo to maintain the study blind.
  Interventions: Biological: CZP 200 mg Q2W; Other: Placebo
- CZP 400 mg Q4W (Experimental): Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 400 mg CZP sc every 4 weeks (Q4W) from Week 8 onwards.
  Subjects received 2 injections of Placebo every 4 weeks in between the 2 injections of 200 mg CZP to maintain the study blind.
  Interventions: Biological: CZP 400 mg Q4W; Other: Placebo
- Placebo (Placebo Comparator): Matching Placebo to CZP injections from Week 0 to Week 24. Placebo subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group on Week 16.
  After 24 weeks, all subjects were randomized to active treatment with CZP 200 mg Q2W or CZP 400 mg Q4W.
  Interventions: Other: Placebo
- Placebo to CZP 200 mg escape on Week 16 (Other): Matching Placebo to CZP injections from Week 0 to Week 16. Subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group on Week 16 and were treated with three loading doses of CZP 400 mg sc on Weeks 16, 18 and 20, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 22 onwards. Additionally, Placebo injections were administered as appropriate in order to maintain the study blind.
  Interventions: Biological: CZP 200 mg Q2W; Other: Placebo
- Placebo to CZP 400 mg escape on Week 16 (Other): Matching Placebo to CZP injections from Week 0 to Week 16. Subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group on Week 16 and were treated with three loading doses of CZP 400 mg sc on Weeks 16, 18 and 20, followed by 400 mg CZP sc every 4 weeks (Q4W) from Week 24 onwards. Additionally, Placebo injections were administered as appropriate in order to maintain the study blind.
  Interventions: Biological: CZP 400 mg Q4W; Other: Placebo
- Placebo to CZP 200 mg on Week 24 (Other): Matching Placebo to CZP injections from Week 0 to Week 24. Three loading doses of CZP 400 mg sc were given on Weeks 24, 26 and 28, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 30 onwards. Additionally, Placebo injections were administered as appropriate in order to maintain the study blind.
  Interventions: Biological: CZP 200 mg Q2W; Other: Placebo
- Placebo to CZP 400 mg on Week 24 (Other): Matching Placebo to CZP injections from Week 0 to Week 24. Three loading doses of CZP 400 mg sc were given on Weeks 24, 26 and 28, followed by 400 mg CZP sc every 4 weeks (Q4W) from Week 32 onwards. Additionally, Placebo injections were administered as appropriate in order to maintain the study blind.
  Interventions: Biological: CZP 400 mg Q4W; Other: Placebo

INTERVENTIONS:
Biological: CZP 200 mg Q2W — 200 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 2 weeks (Q2W).
  Other Names: Cimzia; CZP; Certolizumab Pegol
  Arms: CZP 200 mg Q2W; Placebo to CZP 200 mg escape on Week 16; Placebo to CZP 200 mg on Week 24
Biological: CZP 400 mg Q4W — 400 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 4 weeks (Q4W).
  Other Names: Cimzia; CZP; Certolizumab Pegol
  Arms: CZP 400 mg Q4W; Placebo to CZP 400 mg escape on Week 16; Placebo to CZP 400 mg on Week 24
Other: Placebo — Matching Placebo to CZP injection.

SUMMARY:
The study is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of two dose regimens of Certolizumab Pegol (CZP) in subjects with active axial Spondyloarthritis (axial SpA).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of adult-onset axial Spondyloarthritis (SpA) of at least 3 months' duration as defined by the specified Assessment of Spondyloarthritis International Society (ASAS) criteria
* Active disease as defined by:

  * Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥ 4
  * Back pain ≥ 4 on a 0 to 10 Neurobehavioral Rating Scale (NRS) (from BASDAI item 2)
  * C-Reactive Protein (CRP) > ULN (Upper Limit of Normal) and/or current evidence (ie, within the last 3 months from Screening) for Sacroiliitis on Magnetic Resonance Imaging (MRI) as defined by Assessment of Spondyloarthritis International Society (ASAS) criteria
* Intolerance to or inadequate response to at least 1 Nonsteroidal Anti-Inflammatory Drug (NSAID)

Exclusion Criteria:

* Presence of total Spinal Ankylosis ("bamboo spine")
* Diagnosis of any other Inflammatory Arthritis
* Prior treatment with any experimental biological agents for treatment of Axial Spondyloarthritis (SpA)
* Exposure to more than 1 TNF-antagonist or to more than 2 previous biological agents for Axial Spondyloarthritis (SpA)
* History of or current chronic or recurrent infections
* High risk of infection
* Recent live vaccination
* Concurrent malignancy or a history of malignancy
* Class III or IV congestive heart failure - New York Heart Association (NYHA)
* Demyelinating disease of the central nervous system
* Female subjects who are breastfeeding, pregnant or plan to become pregnant during the study or within 3 months following the last dose of the investigational product
* Subjects with any other condition which, in the investigator's judgment, would make the subject unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 UCB
Locations (104):
- United States (32):
  - 961, Birmingham, Alabama
  - 953, Tuscaloosa, Alabama
  - 954, Peoria, Arizona
  - 971, Scottsdale, Arizona
  - 987, Tucson, Arizona
  - 974, La Jolla, California
  - 973, Los Angeles, California
  - 966, Palm Desert, California
  - 952, San Diego, California
  - 957, Aventura, Florida
  - 962, Fort Lauderdale, Florida
  - 959, Orange Park, Florida
  - 990, Pinellas Park, Florida
  - 958, Vero Beach, Florida
  - 964, Hagerstown, Maryland
  - 969, Eagan, Minnesota
  - 984, Flowood, Mississippi
  - 965, Florissant, Missouri
  - 950, St Louis, Missouri
  - 985, Brooklyn, New York
  - 963, Asheville, North Carolina
  - 977, Cleveland, Ohio
  - 951, Middleburg Heights, Ohio
  - 970, Oklahoma City, Oklahoma
  - 982, Portland, Oregon
  - 972, Duncansville, Pennsylvania
  - 975, Dallas, Texas
  - 978, Houston, Texas
  - 983, Houston, Texas
  - 967, San Antonio, Texas
  - 981, Salt Lake City, Utah
  - 968, Seattle, Washington
- Argentina (9):
  - 700, Buenos Aires
  - 701, Buenos Aires
  - 704, Buenos Aires
  - 705, Córdoba
  - 709, La Plata
  - 706, Rosario
  - 710, San Juan
  - 702, San Miguel de Tucumán
  - 708, San Miguel de Tucumán
- Belgium (3):
  - 153, Brussels
  - 152, Ghent
  - 151, Liège
- Brazil (4):
  - 760, Campinas
  - 750, Curitiba
  - 761, Goiânia
  - 756, São Paulo
- Canada (5):
  - 907, Victoria, British Columbia
  - 903, Winnipeg, Manitoba
  - 900, St. John's, Newfoundland and Labrador
  - 910, Windsor, Ontario
  - 902, Sainte-Foy, Quebec
- Czechia (6):
  - 504, Brno
  - 501, Hlučín
  - 500, Pardubice
  - 502, Prague
  - 505, Terezín
  - 503, Zlín
- France (6):
  - 200, Boulogne-Billan Court
  - 201, Lille
  - 205, Limoges
  - 206, Montpellier
  - 204, Paris
  - 202, Tours
- Germany (9):
  - 257, Berlin
  - 258, Berlin
  - 255, Freiburg im Breisgau
  - 254, Hamburg
  - 250, Herne
  - 253, Leipzig
  - 260, München
  - 263, München
  - 256, Ratingen
- Hungary (5):
  - 303, Budapest
  - 305, Budapest
  - 302, Debrecen
  - 306, Miskolc
  - 300, Veszprém
- Italy (3):
  - 352, Ancona
  - 351, Florence
  - 350, Pisa
- Mexico (2):
  - 802, Cuernavaca
  - 801, Monterrey
- Netherlands (2):
  - 401, Maastricht
  - 400, Rotterdam
- Poland (10):
  - 458, Bialystok
  - 452, Dąbrówka
  - 455, Elblag
  - 459, Gdanks
  - 457, Krakow
  - 450, Lublin
  - 454, Poznan
  - 453, Torun
  - 456, Warsaw
  - 462, Warsaw
- Spain (4):
  - 550, Mérida
  - 554, Santander
  - 552, Santiago de Compostela
  - 553, Seville
- United Kingdom (4):
  - 605, Barnsley
  - 600, Leeds
  - 602, London
  - 601, Salford

REFERENCES:
- [Result] Landewe R, Braun J, Deodhar A, Dougados M, Maksymowych WP, Mease PJ, Reveille JD, Rudwaleit M, van der Heijde D, Stach C, Hoepken B, Fichtner A, Coteur G, de Longueville M, Sieper J. Efficacy of certolizumab pegol on signs and symptoms of axial spondyloarthritis including ankylosing spondylitis: 24-week results of a double-blind randomised placebo-controlled Phase 3 study. Ann Rheum Dis. 2014 Jan;73(1):39-47. doi: 10.1136/annrheumdis-2013-204231. Epub 2013 Sep 6. PMID 24013647
- [Derived] Proft F, Vahldiek JL, Nicolaes J, Tham R, Hoepken B, Ufuktepe B, Poddubnyy D, Bressem KK. Machine learning vs human experts: sacroiliitis analysis from the RAPID-axSpA and C-OPTIMISE phase 3 axSpA trials. Rheumatol Adv Pract. 2025 Apr 18;9(2):rkae118. doi: 10.1093/rap/rkae118. eCollection 2025. PMID 40256636
- [Derived] Rudwaleit M, Marzo-Ortega H, Navarro-Compan V, Tham R, Kumke T, Bauer L, de Peyrecave N, Kim M, Van den Bosch F. Exploratory analysis of the potential disconnect between objective inflammatory response and clinical response following certolizumab pegol treatment in patients with active axial spondyloarthritis. RMD Open. 2024 Aug 28;10(3):e004369. doi: 10.1136/rmdopen-2024-004369. PMID 39209369
- [Derived] Baraliakos X, Kruse S, Auteri SE, de Peyrecave N, Nurminen T, Kumke T, Hoepken B, Braun J. Certolizumab pegol treatment in axial spondyloarthritis mitigates fat lesion development: 4-year post-hoc MRI results from a phase 3 study. Rheumatology (Oxford). 2022 Jul 6;61(7):2875-2885. doi: 10.1093/rheumatology/keab841. PMID 34791107
- [Derived] Landewe R, Nurminen T, Davies O, Baeten D. A single determination of C-reactive protein does not suffice to declare a patient with a diagnosis of axial spondyloarthritis 'CRP-negative'. Arthritis Res Ther. 2018 Sep 14;20(1):209. doi: 10.1186/s13075-018-1707-8. PMID 30217232
- [Derived] van der Heijde D, Braun J, Rudwaleit M, Purcaru O, Kavanaugh AF. Improvements in workplace and household productivity with certolizumab pegol treatment in axial spondyloarthritis: results to week 96 of a phase III study. RMD Open. 2018 Apr 9;4(1):e000659. doi: 10.1136/rmdopen-2018-000659. eCollection 2018. PMID 29670761
- [Derived] van der Heijde D, Baraliakos X, Hermann KA, Landewe RBM, Machado PM, Maksymowych WP, Davies OR, de Peyrecave N, Hoepken B, Bauer L, Nurminen T, Braun J. Limited radiographic progression and sustained reductions in MRI inflammation in patients with axial spondyloarthritis: 4-year imaging outcomes from the RAPID-axSpA phase III randomised trial. Ann Rheum Dis. 2018 May;77(5):699-705. doi: 10.1136/annrheumdis-2017-212377. Epub 2018 Jan 17. PMID 29343510
- [Derived] Braun J, Baraliakos X, Hermann KG, Landewe R, Machado PM, Maksymowych WP, Davies O, Hoepken B, Nurminen T, Stach C, van der Heijde D. Effect of certolizumab pegol over 96 weeks of treatment on inflammation of the spine and sacroiliac joints, as measured by MRI, and the association between clinical and MRI outcomes in patients with axial spondyloarthritis. RMD Open. 2017 Apr 24;3(1):e000430. doi: 10.1136/rmdopen-2017-000430. eCollection 2017. PMID 28848654
- [Derived] van der Heijde D, Dougados M, Landewe R, Sieper J, Maksymowych WP, Rudwaleit M, Van den Bosch F, Braun J, Mease PJ, Kivitz AJ, Walsh J, Davies O, Bauer L, Hoepken B, Peterson L, Deodhar A. Sustained efficacy, safety and patient-reported outcomes of certolizumab pegol in axial spondyloarthritis: 4-year outcomes from RAPID-axSpA. Rheumatology (Oxford). 2017 Sep 1;56(9):1498-1509. doi: 10.1093/rheumatology/kex174. PMID 28498975
- [Derived] van der Heijde D, Deodhar A, Fleischmann R, Mease PJ, Rudwaleit M, Nurminen T, Davies O. Early Disease Activity or Clinical Response as Predictors of Long-Term Outcomes With Certolizumab Pegol in Axial Spondyloarthritis or Psoriatic Arthritis. Arthritis Care Res (Hoboken). 2017 Jul;69(7):1030-1039. doi: 10.1002/acr.23092. Epub 2017 Jun 2. PMID 27696727
- [Derived] Rudwaleit M, Rosenbaum JT, Landewe R, Marzo-Ortega H, Sieper J, van der Heijde D, Davies O, Bartz H, Hoepken B, Nurminen T, Deodhar A. Observed Incidence of Uveitis Following Certolizumab Pegol Treatment in Patients With Axial Spondyloarthritis. Arthritis Care Res (Hoboken). 2016 Jun;68(6):838-44. doi: 10.1002/acr.22848. PMID 26815944
- [Derived] Sieper J, Kivitz A, van Tubergen A, Deodhar A, Coteur G, Woltering F, Landewe R. Impact of Certolizumab Pegol on Patient-Reported Outcomes in Patients With Axial Spondyloarthritis. Arthritis Care Res (Hoboken). 2015 Oct;67(10):1475-80. doi: 10.1002/acr.22594. PMID 25832312
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multicenter study with 128 sites in North America, Latin America, Western Europe, and Central/Eastern Europe. 325 subjects are included in Randomized Set (RS) shown in Participant Flow for the interim period, and 315 for the final analysis (10 subjects dropped out before receiving a CZP dose), which is an Intention-to-Treat (ITT) dataset.
Pre-assignment Details: Patients with positive Tuberculosis (TB) tests within Screening Period, but no signs and symptoms of active TB had to be treated with prophylactic TB treatment for at least 4 weeks prior to first study drug administration.
Groups:
- Placebo: Matching Placebo to Certolizumab Pegol (CZP) injections from Week 0 to Week 24. Placebo subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group on Week 16.
  After 24 weeks, all subjects were randomized to active treatment with CZP 200 mg every two weeks (Q2W) or CZP 400 mg every four weeks (Q4W).
  Placebo : Matching Placebo to CZP injection.
- CZP 200 mg Q2W: Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 onwards.
  At every visit, subjects received one injection of 200 mg CZP and one injection of Placebo to maintain the study blind.
  Placebo : Matching Placebo to CZP injection.
  CZP 200 mg Q2W : 200 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 2 weeks (Q2W).
- CZP 400 mg Q4W: Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 400 mg CZP sc every 4 weeks (Q4W) from Week 8 onwards.
  Subjects received 2 injections of Placebo every 4 weeks in between the 2 injections of 200 mg CZP to maintain the study blind.
  Placebo : Matching Placebo to CZP injection.
  CZP 400 mg Q4W : 400 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 4 weeks (Q4W).
- All CZP 200 mg: All subjects who received CZP at the specified dose (200 mg) at some point during the study, including subjects who were originally randomized to receive placebo and were switched to CZP at Week 16 or Week 24.
  Placebo : Matching Placebo to CZP injection.
  CZP 200 mg Q2W : 200 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 2 weeks (Q2W).
- All CZP 400 mg: All subjects who received CZP at the specified dose (400 mg) at some point during the study, including subjects who were originally randomized to receive placebo and were switched to CZP at Week 16 or Week 24.
  Placebo : Matching Placebo to CZP injection.
  CZP 400 mg Q4W : 400 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 4 weeks (Q4W).
Period: Double Blind Period (Weeks 0-24)
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q4W | All CZP 200 mg | All CZP 400 mg
Started | 107 (Completed 24-weeks Double-blind Period) | 111 (Completed 24-weeks Double-blind Period) | 107 (Completed 24-weeks Double-blind Period) | 0 | 0
Completed | 95 | 105 | 98 | 0 | 0
Not Completed | 12 | 6 | 9 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 3 | 0 | 0
Not completed — Protocol Violation | 6 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 0
Not completed — SAE, non-fatal | 2 | 2 | 3 | 0 | 0
Period: Open-Label Period (Weeks 48-204)
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q4W | All CZP 200 mg | All CZP 400 mg
Started | 0 | 0 | 0 | 158 | 157
Completed | 0 | 0 | 0 | 99 | 100
Not Completed | 0 | 0 | 0 | 59 | 57
Not completed — Lack of Efficacy | 0 | 0 | 0 | 4 | 14
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 22 | 15
Not completed — Other | 0 | 0 | 0 | 2 | 4
Not completed — SAE, non-fatal | 0 | 0 | 0 | 7 | 4
Not completed — AE, non-serious non-fatal | 0 | 0 | 0 | 16 | 13
Not completed — SAE, non-fatal + AE, non-serious/fatal | 0 | 0 | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS), which is an Intention-to-Treat (ITT) dataset.
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q4W | Total Title
Number analyzed (Participants) | 107 | 111 | 107 | 325
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 102 | 110 | 105 | 317
  >=65 years | 5 | 1 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean age | 39.9 (12.4) | 39.1 (11.9) | 39.8 (39.9) | 39.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 39 | 125
  Male | 65 | 67 | 68 | 200
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 82.142 (18.147) | 79.305 (18.599) | 83.893 (18.855) | 81.757 (18.576)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.704 (9.692) | 171.769 (10.171) | 172.753 (9.607) | 171.739 (9.834)

OUTCOME MEASURES:

1. Primary Outcome: Assessment in Axial Spondyloarthritis International Society 20 % (ASAS20) Response Criteria at Week 12
Description: The ASAS20 is defined as an improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 following domains:
  * Patient's Global Assessment of Disease Activity
  * Pain assessment (total spinal pain)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration)
  and absence of deterioration in the potential remaining domain (deterioration is defined as a relative worsening of at least 20 % and an absolute worsening of at least 1 unit).
Time Frame: Week 12
Population: Intention-to-treat dataset was the Randomized Set (RS). RS with non-responder imputation: subjects who withdrew for any reason or placebo subjects who used escape medication are considered as non-responders from drop out timepoint or when escape therapy was initiated. Subjects with missing data at a visit are non-responders for that visit, too.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo (FAS): Matching Placebo to Certolizumab Pegol (CZP) injections from Week 0 to Week 24. Placebo subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group on Week 16.
  After 24 weeks, all subjects were randomized to active treatment with CZP 200 mg every two weeks (Q2W) or CZP 400 mg every four weeks (Q4W).
  Placebo : Matching Placebo to CZP injection.
- CZP 200 mg Q2W (FAS): Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 onwards.
  At every visit, subjects received one injection of 200 mg CZP and one injection of Placebo to maintain the study blind.
  Placebo : Matching Placebo to CZP injection.
  CZP 200 mg Q2W : 200 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 2 weeks (Q2W).
- CZP 400 mg Q4W (FAS): Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 400 mg CZP sc every 4 weeks (Q4W) from Week 8 onwards.
  Subjects received 2 injections of Placebo every 4 weeks in between the 2 injections of 200 mg CZP to maintain the study blind.
  Placebo : Matching Placebo to CZP injection.
  CZP 400 mg Q4W : 400 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 4 weeks (Q4W).
- CZP 200 mg Q2W and CZP 400 mg Q4W (FAS): This arm shows a combination of arm CZP 200 mg Q2W and arm CZP 400 mg Q4W. Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W)/ 400 mg CZP sc every 4 weeks (Q4W) from Week 6/ Week 8 onwards.
  Subjects in both CZP arms received additional placebo injections to maintain the study blind.
  Placebo : Matching Placebo to CZP injection.
  CZP 200 mg Q2W : 200 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 2 weeks (Q2W).
  CZP 400 mg Q4W : 400 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 4 weeks (Q4W).
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 107 | 111 | 107 | 218
percentage of participants | 38.3 [29.1 to 47.5] | 57.7 [48.5 to 66.8] | 63.6 [54.4 to 72.7] | 60.6 [54.1 to 67.0]
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); A hierarchical test procedure was applied to protect the overall significance level for the multiplicity of dose groups and endpoints. Conditional on the first test being significant, the second hypothesis was tested with the same alpha level of 5 %. Statistical testing for the following hypotheses was performed only if the previous null hypothesis in the hierarchy was rejected; Test type: Superiority or Other; p = 0.004, Wald-test, 2-sided — Difference of Certolizumab Pegol 200 mg versus Placebo (and corresponding 95 % Confidence Interval and p-value) were estimated using a standard two-sided Wald asymptotic test with a 5 % alpha level; Wald test and Confidence Interval (CI) calculation were performed without continuity correction; Mean Difference (Final Values) = 19.3, 95% CI 2-sided [6.3 to 32.4]
Statistical Analysis 2: Comparison: Placebo (FAS) vs CZP 400 mg Q4W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald-test, 2-sided — Difference of Certolizumab Pegol 400 mg versus Placebo (and corresponding 95 % Confidence Interval and p-value) were estimated using a standard two-sided Wald asymptotic test with a 5 % alpha level; Wald test and Confidence Interval (CI) calculation were performed without continuity correction; Mean Difference (Final Values) = 25.2, 95% CI 2-sided [12.3 to 38.2]

2. Secondary Outcome: Assessment in Axial Spondyloarthritis International Society 20 % (ASAS20) Response Criteria at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 107 | 111 | 107 | 218
percentage of participants | 29.0 [20.4 to 37.6] | 66.7 [57.9 to 75.4] | 70.1 [61.4 to 78.8] | 68.3 [62.2 to 74.5]
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald-test, 2-sided — [p-value comment as in outcome 1, analysis 1]; Wald test and Confidence Interval (CI) calculation were performed without continuity correction; Mean Difference (Final Values) = 37.7, 95% CI 2-sided [25.4 to 50.0]
Statistical Analysis 2: Comparison: Placebo (FAS) vs CZP 400 mg Q4W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald-test, 2-sided — [p-value comment as in outcome 1, analysis 2]; Wald test and Confidence Interval (CI) calculation were performed without continuity correction; Mean Difference (Final Values) = 41.1, 95% CI 2-sided [28.9 to 53.3]

3. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 12
Description: The BASFI assesses physical function in comprising 10 items relating to activities during the past week. Each item ranges from 0 ("Easy") to 10 ("Impossible"). The BASFI is the mean of the 10 scores such that the total score ranges from 0 to 10, with lower scores indicating better physical function. A negative value in BASFI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: From Baseline to Week 12
Population: Intention-to-treat dataset was the Randomized Set (RS). RS with Last Observation Carried Forward (LOCF): for subjects who withdrew for any reason, or subjects with missing Week 12 measurements, last observation prior to the early withdrawal or Week 12 is carried forward to Week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 107 | 111 | 107 | 218
units on a scale | -0.53 [-0.96 to -0.10] | -2.01 [-2.48 to -1.55] | -2.02 [-2.50 to -1.55] | -2.02 [-2.40 to -1.63]
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W and CZP 400 mg Q4W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Difference of CZP 200 mg + 400 mg vs. Placebo was estimated using an ANCOVA model with treatment, region, modified New York criteria and prior TNF-antagonist exposure as factors and Baseline BASFI score as a covariate; Mean Difference (Final Values) = -1.49, 95% CI 2-sided [-1.96 to -1.01], Standard Error of Mean 0.24

4. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 24
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: Intention-to-treat dataset was the Randomized Set (RS). RS with Last Observation Carried Forward (LOCF): for subjects who withdrew for any reason, or subjects with missing Week 24 measurements, or placebo subjects who used escape medication, last observation prior to early withdrawal or Week 24 or before receiving CZP is carried forward to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 107 | 111 | 107 | 218
units on a scale | -0.40 [-0.85 to 0.06] | -2.36 [-2.85 to -1.87] | -2.20 [-2.70 to -1.70] | -2.28 [-2.68 to -1.87]
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W and CZP 400 mg Q4W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-2.38 to -1.38], Standard Error of Mean 0.25

5. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 12
Description: The BASDAI is a validated self-reported instrument which consists of six 10 unit horizontal Numerical Rating Scales (NRSs) to measure severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration, respectively) over the last week. The final BASDAI score ranges from 0 to 10, with lower scores indicating lower disease activity. A negative value in BASDAI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: From Baseline to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 107 | 111 | 107 | 218
units on a scale | -1.22 [-1.65 to -0.78] | -2.82 [-3.29 to -2.35] | -2.80 [-3.28 to -2.33] | -2.81 [-3.20 to -2.43]
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W and CZP 400 mg Q4W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Difference of CZP 200 mg + 400 mg vs. Placebo was estimated using an ANCOVA model with treatment, region, modified New York criteria and prior TNF-antagonist exposure as factors and Baseline BASDAI score as a covariate; Mean Difference (Final Values) = -1.60, 95% CI 2-sided [-2.07 to -1.12], Standard Error of Mean 0.24

6. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 24
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 107 | 111 | 107 | 218
units on a scale | -1.05 [-1.50 to -0.60] | -3.08 [-3.57 to -2.60] | -3.01 [-3.50 to -2.52] | -3.05 [-3.45 to -2.65]
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W and CZP 400 mg Q4W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-2.49 to -1.50], Standard Error of Mean 0.25

7. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 12
Description: The BASMI characterizes the spinal mobility of subjects with axial Spondyloarthritis (SpA) and Ankylosing Spondylitis (AS). It is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 is calculated for each item based on the measurement. The mean of the sum of the 5 scores provides the BASMI score. The higher the BASMI score the more severe the patient's limitation of movement due to their axial SpA. A negative value in BASMI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: From Baseline to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 107 | 111 | 107 | 218
units on a scale | -0.13 [-0.31 to 0.05] | -0.60 [-0.79 to -0.40] | -0.46 [-0.66 to -0.26] | -0.53 [-0.69 to -0.37]
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W and CZP 400 mg Q4W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Difference of CZP 200 mg + 400 mg vs. Placebo was estimated using an ANCOVA model with treatment, region, modified New York criteria and prior TNF-antagonist exposure as factors and Baseline BASMI score as a covariate; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.60 to -0.20], Standard Error of Mean 0.10

8. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 24
Description: The BASMI characterizes the spinal mobility of subjects with axial SpA and AS. It is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 is calculated for each item based on the measurement. The mean of the sum of the 5 scores provides the BASMI score. The higher the BASMI score the more severe the patient's limitation of movement due to their axial SpA. A negative value in BASMI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: From Baseline to Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 107 | 111 | 107 | 218
units on a scale | -0.07 [-0.27 to 0.12] | -0.54 [-0.75 to -0.34] | -0.49 [-0.70 to -0.28] | -0.52 [-0.69 to -0.34]
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W and CZP 400 mg Q4W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.66 to -0.23], Standard Error of Mean 0.11

9. Secondary Outcome: Change From Baseline in the Spine Ankylosing Spondylitis Spine Magnetic Resonance Imaging (MRI) Scoring System for Disease Activity (ASspiMRI-a) in the Berlin Modification at Week 12
Description: The Berlin modification of the ASspiMRI-a is a scoring system with a concentration on Short-Tau-Inversion Recovery (STIR) sequences without other fat saturation techniques. It quantifies changes in 23 Vertebral Units (VU) of the spine. A VU is defined as the region between 2 virtual lines through the middle of each vertebra. Active inflammation is scored by grading the degree of bone marrow edema from 0 to 3 in 1 dimension on 1 or more consecutive slices that represent the highest level of inflammation in a particular VU. Total spine ASspiMRI-a score in the Berlin modification can range from 0 to 69 with higher scores indicating higher disease activity. A negative value in total spine ASspiMRI-a score change from Baseline indicates an improvement from Baseline. The higher the negative value the higher the reduction of inflammation.
Time Frame: From Baseline to Week 12
Population: The analysis was performed in the Magnetic Resonance Imaging (MRI) Set, a subgroup of subjects participating in an imaging substudy, where MRI measurements at Baseline and Week 12 were performed. Of the 325 patients randomized, 153 participated in the imaging substudy. Of these 153 subjects in the MRI Set, 148 are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 49 | 47 | 52 | 99
units on a scale | 0.39 (4.04) | -3.39 (5.59) | -2.16 (3.61) | -2.74 (4.67)

10. Secondary Outcome: Change From Baseline in Sacroiliac Spondyloarthritis Research Consortium of Canada (SPARCC) Score at Week 12
Description: The SPARCC scoring method for lesions found on the Magnetic Resonance Imaging (MRI) is based on an abnormal increased signal on the Short-Tau-Inversion Recovery (STIR) sequence, representing bone marrow edema. Total Sacroiliac (SI) joint SPARCC score can range from 0 to 72 with higher scores indicating higher joint inflammation. A negative value in SPARCC change from Baseline indicates an improvement from Baseline. The higher the negative value the higher the reduction of inflammation.
Time Frame: From Baseline to Week 12
Population: The analysis was performed in the Magnetic Resonance Imaging (MRI) Set, a subgroup of subjects participating in an imaging substudy, where MRI measurements at Baseline and Week 12 were performed. Of the 325 patients randomized, 153 participated in the imaging substudy. Of these 153 subjects in the MRI Set, 140 are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q4W (FAS) | CZP 200 mg Q2W and CZP 400 mg Q4W (FAS)
Number analyzed (Participants) | 45 | 45 | 50 | 95
units on a scale | -1.33 (8.33) | -3.61 (6.94) | -4.98 (8.47) | -4.33 (7.77)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Baseline (Week 0) until study end (Week 204). AEs refer to the Safety Set including all randomized subjects who took at least 1 dose of CZP.
Description: As per study design, placebo arm subjects shifted either at Week 16 or 24 to CZP treatment. For the Placebo (PBO) group, CZP data from PBO subjects are not utilized. The All CZP 200 mg + 400 mg group shows CZP 200 mg, CZP 400 mg and the escaped PBO subjects with their CZP data.
Groups:
- All CZP 200 mg (Safety Analysis): All subjects who received CZP at the specified dose (200 mg) at some point during the study, including subjects who were originally randomized to receive placebo and were switched to CZP at Week 16 or Week 24.
  Placebo : Matching Placebo to CZP injection.
  CZP 200 mg Q2W : 200 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 2 weeks (Q2W).
- All CZP 400 mg (Safety Analysis): All subjects who received CZP at the specified dose (400 mg) at some point during the study, including subjects who were originally randomized to receive placebo and were switched to CZP at Week 16 or Week 24.
  Placebo : Matching Placebo to CZP injection.
  CZP 400 mg Q4W : 400 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 4 weeks (Q4W).
- All CZP 200 mg + 400 mg: This arm shows all patients treated with Certolizumab Pegol (CZP) at least once. Hence, this arm is a combination of arm All CZP 200 mg and arm All CZP 400 mg.
Arm/Group | All CZP 200 mg (Safety Analysis) | All CZP 400 mg (Safety Analysis) | All CZP 200 mg + 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 35/158 | 34/157 | 69/315 | 5/107
Other Adverse Events (participants affected / at risk) | 142/158 | 127/157 | 269/315 | 28/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All CZP 200 mg (Safety Analysis) (N=158) | All CZP 400 mg (Safety Analysis) (N=157) | All CZP 200 mg + 400 mg (N=315) | Placebo (N=107)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sigmoiditis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Cholelithiasis migration (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mycobacterial infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (5) | 0 (0) | 3 (5) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Latent tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholesterol granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Squamous cell carcinoma of the (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (2) | 1 (1) | 2 (3) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bone graft (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All CZP 200 mg (Safety Analysis) (N=158) | All CZP 400 mg (Safety Analysis) (N=157) | All CZP 200 mg + 400 mg (N=315) | Placebo (N=107)
Uveitis (Eye disorders) | 11 (15) | 8 (12) | 19 (27) | 0 (0)
Conjunctivitis (Eye disorders) | 5 (6) | 8 (9) | 13 (15) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (13) | 20 (26) | 30 (39) | 0 (0)
Gastritis (Gastrointestinal disorders) | 8 (8) | 5 (5) | 13 (13) | 0 (0)
Seasonal allergy (Immune system disorders) | 7 (8) | 8 (11) | 15 (19) | 0 (0)
Nasopharyngitis (Infections and infestations) | 47 (80) | 43 (83) | 90 (163) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 35 (53) | 28 (58) | 63 (111) | 3 (3)
Bronchitis (Infections and infestations) | 24 (28) | 17 (18) | 41 (46) | 0 (0)
Pharyngitis (Infections and infestations) | 24 (36) | 11 (17) | 35 (53) | 0 (0)
Sinusitis (Infections and infestations) | 17 (21) | 8 (10) | 25 (31) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (17) | 11 (15) | 21 (32) | 4 (4)
Rhinitis (Infections and infestations) | 15 (22) | 6 (8) | 21 (30) | 0 (0)
Influenza (Infections and infestations) | 9 (10) | 11 (14) | 20 (24) | 0 (0)
Tonsillitis (Infections and infestations) | 8 (10) | 9 (11) | 17 (21) | 0 (0)
Oral herpes (Infections and infestations) | 9 (23) | 6 (7) | 15 (30) | 0 (0)
Cystitis (Infections and infestations) | 8 (13) | 6 (10) | 14 (21) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 9 (9) | 14 (14) | 0 (0)
Viral infection (Infections and infestations) | 9 (10) | 4 (4) | 13 (14) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 10 (18) | 9 (11) | 19 (29) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 14 (16) | 17 (23) | 31 (39) | 2 (3)
Alanine aminotransferase increased (Investigations) | 11 (14) | 8 (10) | 19 (24) | 0 (0)
Tuberculin test positive (Investigations) | 8 (8) | 7 (7) | 15 (15) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 8 (9) | 14 (15) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (42) | 11 (20) | 33 (62) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (18) | 11 (19) | 25 (37) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 12 (22) | 13 (14) | 25 (36) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 11 (17) | 5 (8) | 16 (25) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (11) | 3 (4) | 13 (15) | 0 (0)
Headache (Nervous system disorders) | 17 (25) | 18 (31) | 35 (56) | 7 (11)
Depression (Psychiatric disorders) | 9 (10) | 4 (5) | 13 (15) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 11 (13) | 24 (29) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 6 (6) | 18 (21) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 11 (15) | 14 (18) | 25 (33) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 8 (14) | 6 (9) | 14 (23) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 4 (6) | 8 (13) | 12 (19) | 0 (0)
Hypertension (Vascular disorders) | 20 (26) | 11 (11) | 31 (37) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days